CLINICAL TRIAL: NCT03673228
Title: Preventing Smoking Relapse After Total Joint Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-00723
Record Dates: First submitted 2018-08-27; First posted 2018-09-17 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the Intervention Arm will receive counseling that includes:
  * A Visit prior to discharge
  * Follow up calls after discharge
  * Text Messaging Support
  * Caregiver Support
  Interventions: Behavioral: Comprehensive Relapse Prevention Intervention; Drug: Nicotine Replacement Therapy (NRT)
- Standard treatment (Active Comparator): Patients will receive current usual care.
  Interventions: Behavioral: Standard Treatment Counseling; Drug: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Behavioral: Comprehensive Relapse Prevention Intervention — This intervention consists of 4 components:
  1. Visit Prior to Discharge: counselor from research team will visit patient at hospital bedside to provide counseling
  2. Follow up calls after discharge: 6 proactive counseling calls and initiate unlimited reactive calls to their counselor, at days 1,3,7,14,30,an 60 days after hospital visit
  3. Text messaging support: patients will be registered in NCI's Smokefree TXT while in the hospital and will receive multiple daily messages, designed for someone who has already quit
  4. Caregiver support: 10 minute training session to the caregiver on how to help patient prevent relapse by increasing self efficacy, maintaining motivation and dealing with high risk situations
  Arms: Intervention Group
Behavioral: Standard Treatment Counseling — Participants will receive two 10 minute counseling calls from the staff of the preoperative counseling program during the first month after the hospital discharge
  Arms: Standard treatment
Drug: Nicotine Replacement Therapy (NRT) — Patients in both arms will be encouraged to receive NRT

SUMMARY:
Hospitalization for elective knee or hip replacement surgery presents an outstanding opportunity to motivate people to quit smoking, because it provides an opportunity to encourage patients to remain smoke-free as they proactively quit to optimize their surgery outcomes. This study will conduct a comparative effectiveness trial of patients who quit smoking pre-operatively, comparing the current standard of care with a novel comprehensive relapse prevention intervention guided by Marlatt's Relapse Prevention Model.

DETAILED DESCRIPTION:
The specific aims of this study are to evaluate the effectiveness and cost-effectiveness of the relapse prevention intervention and will: 1) compare the effectiveness of standard post-operative cessation treatment with a comprehensive relapse prevention intervention on smoking cessation outcomes; 2) conduct a comparative economic analysis to assess the value of the relapse prevention intervention for patients and the healthcare system; and 3) explore the impact of the interventions on surgical complications and readmissions.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants

* Received preoperative smoking cessation counseling through Orthopedic Surgery Quit Smoking Program
* Undergoing elective knee or hip arthroplasty surgery
* Have not smoked any cigarettes in the week prior to admission and carbon monoxide 4 ppm46,47
* Have a cell phone (for text messaging)
* Provide informed consent in English

Caregiver participants:

* Age ≥ 18 years
* Be a caregiver of the patient participant
* Provide informed consent in English

Exclusion Criteria:

* Patients will be excluded if they used smokeless tobacco or an electronic cigarette in the last 30 days.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Self Reported Relapse Rate for Usual Care Arm | 3 Months
  Measured using the modified Dillman method
Self Reported Relapse Rate for Usual Care Arm | 6 Months
  Measured using the modified Dillman method
Self Reported Relapse Rate for Usual Care Arm | 12 Months
  Measured using the modified Dillman method
Self Reported Relapse Rate for relapse prevention intervention arm | 3 Months
  Measured using the modified Dillman method
Self Reported Relapse Rate for relapse prevention intervention arm | 6 Months
  Measured using the modified Dillman method
Self Reported Relapse Rate for relapse prevention intervention arm | 12 Months
  Measured using the modified Dillman method

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sherman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided